CLINICAL TRIAL: NCT00224081
Title: Dialysis Patients' Response to IV Iron With Elevated Ferritin
Brief Title: DRIVE Trial (Dialysis Patients' Response to Intravenous [IV] Iron With Elevated Ferritin)
Acronym: DRIVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FER0401
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Anemia, Iron-Deficiency; Kidney Failure, Chronic; Hemodialysis
Keywords: iron deficiency anemia; ferritin; hemodialysis; sodium ferric gluconate; epoetin alfa
MeSH Terms: conditions — Anemia, Iron-Deficiency; Kidney Failure, Chronic | interventions — ferric gluconate

ARMS (2):
- Ferric gluconate (Experimental)
  Interventions: Drug: Sodium ferric gluconate,
- standard of care (No Intervention)

INTERVENTIONS:
Drug: Sodium ferric gluconate, — Sodium ferric gluconate, 125 mg IV given at 8 consecutive hemodialysis sessions
  Arms: Ferric gluconate

SUMMARY:
This study explores the safety and efficacy of intravenous iron therapy in anemic hemodialysis patients treated with epoetin alfa, who have higher serum ferritin levels, but low to normal transferrin saturation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis
* Elevated serum ferritin with low to normal transferrin saturation (TSAT)
* Moderate to severe anemia
* Receiving epoetin alfa treatment

Exclusion Criteria:

* Known sensitivity to Ferrlecit®
* Medical conditions that would confound the efficacy evaluation
* Recent blood transfusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2004-09; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin and anemia medications | 6 weeks

SECONDARY OUTCOMES:
Change in various iron indices | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adel R. Rizkala, Pharm.D., MS, Study Director — Watson Laboratories, Inc.
Locations (29):
- United States (29):
  - Bakersfield, California
  - Glendale, California
  - Los Angeles, California
  - Santa Rosa, California
  - Torrance, California
  - Lauderdale Lakes, Florida
  - Tampa, Florida
  - Roswell, Georgia
  - Waycross, Georgia
  - Crestwood, Illinois
  - Wichita, Kansas
  - Shreveport, Louisiana
  - Boston, Massachusetts
  - Kalamazoo, Michigan
  - Royal Oak, Michigan
  - Columbia, Missouri
  - St Louis, Missouri
  - North Brunswick, New Jersey
  - Brooklyn, New York
  - Minneola, New York
  - New York, New York
  - Youngstown, Ohio
  - Philadelphia, Pennsylvania
  - Chattanooga, Tennessee
  - Knoxville, Tennessee
  - Arlington, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Morgantown, West Virginia

REFERENCES:
- [Result] Coyne DW, Kapoian T, Suki W, Singh AK, Moran JE, Dahl NV, Rizkala AR; DRIVE Study Group. Ferric gluconate is highly efficacious in anemic hemodialysis patients with high serum ferritin and low transferrin saturation: results of the Dialysis Patients' Response to IV Iron with Elevated Ferritin (DRIVE) Study. J Am Soc Nephrol. 2007 Mar;18(3):975-84. doi: 10.1681/ASN.2006091034. Epub 2007 Jan 31. PMID 17267740
- [Result] Singh AK, Coyne DW, Shapiro W, Rizkala AR; DRIVE Study Group. Predictors of the response to treatment in anemic hemodialysis patients with high serum ferritin and low transferrin saturation. Kidney Int. 2007 Jun;71(11):1163-71. doi: 10.1038/sj.ki.5002223. Epub 2007 Mar 28. PMID 17396118
- [Result] Kapoian T, O'Mara NB, Singh AK, Moran J, Rizkala AR, Geronemus R, Kopelman RC, Dahl NV, Coyne DW. Ferric gluconate reduces epoetin requirements in hemodialysis patients with elevated ferritin. J Am Soc Nephrol. 2008 Feb;19(2):372-9. doi: 10.1681/ASN.2007050606. Epub 2008 Jan 23. PMID 18216316
- [Result] Pizzi LT, Bunz TJ, Coyne DW, Goldfarb DS, Singh AK. Ferric gluconate treatment provides cost savings in patients with high ferritin and low transferrin saturation. Kidney Int. 2008 Dec;74(12):1588-95. doi: 10.1038/ki.2008.489. Epub 2008 Oct 1. PMID 19034302